CLINICAL TRIAL: NCT06129604
Title: A Phase 2 Pilot Window of Opportunity Study of the EP2 and EP4 Receptors Inhibitor TPST-1495 in Patients With Endometrial Cancer or Colorectal Cancer Planning to Undergo Surgical Therapy
Brief Title: Pilot Window of Opportunity Trial (POET)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OU-SCC-POET
Record Dates: First submitted 2023-10-02; First posted 2023-11-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Carcinoma (CRC); Endometrial Carcinoma (EC)
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms

STUDY DESIGN:
Intervention Model Description: This pilot window of opportunity study proposes to evaluate the safety and biological efficacy of 50mg TPST-1495 in patients with EC or CRC undergoing surgical therapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- pilot window of opportunity trial of TPST-1495 (Experimental)
  Interventions: Drug: TPST-1495

INTERVENTIONS:
Drug: TPST-1495 — Eligible subjects will receive study treatment of 50mg TPST-1495 taken orally, once a day for 7 days prior and discontinued 3 days prior to scheduled surgery.

SUMMARY:
The proposed clinical trial with TPST-1495 can help people with two types of cancer, Endometrial Cancer (EC) and Colorectal Carcinoma (CRC), who need surgery. The investigator plans to evaluate how well TPST-1495 works against these cancers by checking blood samples and tumor tissues taken before and after the treatment to see if it is an effective treatment option to help the immune system fight against cancer.

DETAILED DESCRIPTION:
TPST-1495, a dual antagonist targeting human prostaglandin E2 receptor subtypes EP2 and EP4, has shown promising safety and possesses potential immunomodulatory and antineoplastic properties in preclinical research. Based on previous clinical research, the investigator proposes that TPST-1495 treatment could offer anti-cancer benefits to endometrial cancer (EC) and colorectal cancer (CRC) patients.

This pilot window-of-opportunity study aims to assess the safety and biological effectiveness of administering 50mg TPST-1495 orally once daily for seven days, with discontinuation three days prior to surgical therapy, involving 10 evaluable patients, with five each from the EC and CRC groups, for a maximum total of 20 participants enrolled to ensure 10 evaluable patients.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent signed and dated by the patient prior to the performance of any study- specific procedures.
2. At least 18 years of age at the time of signature of the informed consent form (ICF)
3. Histologically confirmed endometrial cancer or colorectal cancer of any stage; either newly diagnosed or recurrent cancer, however no prior chemotherapy or radiation will be allowed.
4. Must be candidates for surgical therapy.
5. Male or female patients. Male patients with female partners of childbearing potential and female patients of childbearing potential are required to use two highly effective methods of contraception during the study treatment and for 3 months after the treatment termination visit. In addition, women of childbearing potential are required to undergo serum pregnancy testing at screening, and at the treatment termination visit.

   Male study participants should refrain from sperm donation during study treatment and up to 3 months following the last dose of TPST-1495
6. To have archival tumor tissue specimen available. Otherwise, patients should agree to have tumor biopsy to obtain sufficient tissue for histological assessment.
7. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1.
8. Life expectancy estimated to be > 12 weeks.
9. Adequate organ and marrow function as defined in protocol.

Exclusion Criteria:

1. Concurrent enrollment in another clinical study, unless it is an observational clinical study, a specimen-collection study, or the follow-up period of an interventional study.
2. Patients who used NSAID or COX-2 inhibitors with duration of 4 days or longer within 2 weeks prior to study treatment initiation.
3. Patients with past medical history (PMH) of allergy or hypersensitivity, GI bleed, or ulceration secondary to NSAID's or COX-2 inhibitors.
4. PMH of GI ulcer within one year of treatment initiation or history of untreated helicobacter's pylori infection. Subjects with history of treated helicobacter's pylori infection with confirmation of eradication are eligible.
5. PMH of diverticulitis or any GI bleed within 2 years of treatment initiation.
6. Heart failure is classified by New York Heart Association as Classification II, III or IV.
7. Patients with history of MI or TIA/CVA will be excluded.
8. Active autoimmune disease or inflammatory disorders including inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease) requiring systemic treatment (i.e., with use of disease modifying agents, systemic corticosteroids, or immunosuppressive drug) within 2 years prior to treatment initiation.
9. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations including a history of substance abuse that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
10. Subjects who are receiving anticoagulant therapy or considered to be at increased risk of bleeding (i.e., bleeding disorder or coagulopathy).
11. Psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol and/or follow-up procedures outlined in the protocol.
12. Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen should be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-08-22 (Actual); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
EP2 and EP4 receptor subtypes blood biomarker expression within the PGE2 signaling pathway. | 1 years
  Blood samples from patients with EC and/or CRC will be assessed at screening(pre-dose) and post-surgery to evaluate the expression of EP2 and EP4 receptor biomarkers within the PGE2 signaling pathway, providing insights into impact of TPST-1495 on pharmacodynamic pathway changes.
EP2 and EP4 receptor subtypes tumor biomarker expression within the PGE2 signaling pathway. | 1 years
  Tumor samples from patient with EC and/or CRC will be assessed at screening (pre-dose) and post-surgery to evaluate the expression of EP2 and EP4 receptor biomarkers within the PGE2 signaling pathway, providing insights into impact of TPST-1495 on pharmacodynamic pathway changes.

SECONDARY OUTCOMES:
Antitumor Activity | 2 years
  Number and percentage of participants with EC and/or CRC will be reported for anti-tumor activity of TPST-1495's, based on the measurement involving mean or median values of circulatory immune cells in blood samples and tumor tissues at screening(pre-dose) and post-surgery.
Biological Efficacy | 2 years
  Number and percentage of participants with EC and/or CRC will be assessed for biological efficacy of TPST-1495's, based on the measurement involving mean or median values of circulatory immune cells in blood samples and tumor tissues at screening (pre-dose) and post-surgery.
Rate of dynamic changes in immune cells | 2 years
  This measure involves comparing the mean or median values of pre-blood and post-blood samples to assess the dynamic changes in immune cell populations. Flow cytometry will be utilized to examine alterations in immune cell composition following treatment.
Rate of dynamic Changes in Inflammatory Cytokines and Chemokines | 2 years
  This outcome measure focuses on comparing the mean or median values of pre-blood and post-blood samples to evaluate dynamic changes in inflammatory cytokines and chemokines. Flow cytometry will be employed to assess variations in the levels of these important biomolecules in response to treatment.
Incidences of TPST-1495 drug therapy based potential adverse events | 2 years
  It utilizes CTCAE v5.0 to systematically report and assess the incidence and the severity of potential adverse events that patients may experience during treatment, ensuring consistent and reliable safety assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Susanna Ulahannan, MD, Principal Investigator — OU Health Stephenson Cancer Center
Locations (1):
- OU Health Stephenson Cancer Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No